CLINICAL TRIAL: NCT02454569
Title: Vicente Ferrer HIV Cohort Study
Acronym: VFHCS
Status: Recruiting | Type: Observational
Sponsor: Rural Development Trust Hospital (Other)
Responsible Party: Principal Investigator, Gerardo Alvarez-Uria, Head of the Department of Infectious Diseases, Rural Development Trust Hospital
Other Study IDs: VFHCS
Record Dates: First submitted 2015-05-15; First posted 2015-05-27 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: HIV; Tuberculosis; Cryptococcosis; Opportunistic Infections; Noncommunicable Diseases
MeSH Terms: conditions — Tuberculosis; Cryptococcosis; Opportunistic Infections; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The VFHCS is a long-term prospective cohort study of HIV infected patients from a resource-poor rural setting in India. The aim of the study is to use data collected from routine clinical care in order to describe the epidemiology of HIV and its related conditions in the investigators area, and to study the effectiveness of health interventions in a "real-world" setting (implementation and operational research).

DETAILED DESCRIPTION:
Andhra Pradesh is the state with highest burden of HIV in India. Anantapur is a district situated in the South border of Andhra Pradesh with 72% rural population and adult literacy rate of 74.1% in men and 54.3% in women. In Anantapur, the HIV epidemic is largely driven by heterosexual transmission and it is characterized by poor socioeconomic conditions and high levels of illiteracy.

Rural Development Trust (RDT) is a nongovernmental organization, which provides medical care to people living with HIV free of charge, including medicines, consultation and admission charges. In Bathalapalli Hospital, outpatient clinics and 71 beds are allocated exclusively for HIV or tuberculosis infected patients.

The Vicente Ferrer HIV Cohort Study (VFHCS) is a prospective open cohort study of all HIV infected patients who have attended Bathalapalli RDT Hospital. Routine clinical data from patients are collected prospectively since September 2009 and entered in a SQL-server database using C# as front end. Details of route of transmission, HIV associated risk factors and socio-demographic data are collected at enrolment. Data collected include medical treatment (antiretroviral treatment and other medications), laboratory investigations (haemogram, renal function tests, liver function tests, CD4 lymphocyte count, bacterial infections), and standardized diagnoses.

The objective of the VFHCS is to describe social and medical aspects related to HIV in the investigators setting, including:

1. Epidemiology: trends in HIV incidence, transmission mechanisms, socioeconomic risk factors associated with HIV.
2. Incidence and prevalence of opportunistic infections, especially tuberculosis and cryptococcosis.
3. Life expectancy and factors associated with mortality
4. Describe the retention across the continuum of care and investigate factors associated with loss to follow-up.
5. Toxicity and effectiveness of antiretroviral therapy.
6. Effectiveness of programmes to prevent mother to child transmission.
7. Incidence and prevalence of non-communicable diseases such as cancer or cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Positive serology for HIV

Exclusion Criteria:

* Refuse to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV infected patients
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2009-09; Primary Completion 2039-09 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | Time to event methods will be used. Participants will be followed from HIV diagnosis until death, assessed up to 30 years
  Survival since diagnosis of HIV infection

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Alvarez-Uria, Principal Investigator — Rural Development Trust
Locations (1):
- RDT Hospital, Battalapalli, Andhra Pradesh, India

REFERENCES:
- [Result] Alvarez-Uria G, Midde M, Pakam R, Naik PK. Gender differences, routes of transmission, socio-demographic characteristics and prevalence of HIV related infections of adults and children in an HIV cohort from a rural district of India. Infect Dis Rep. 2012 Feb 17;4(1):e19. doi: 10.4081/idr.2012.e19. eCollection 2012 Jan 2. PMID 24470926
- [Result] Alvarez-Uria G, Naik PK, Pakam R, Midde M. Early HIV viral load determination after initiating first-line antiretroviral therapy for indentifying patients with high risk of developing virological failure: data from a cohort study in a resource-limited setting. Trop Med Int Health. 2012 Sep;17(9):1152-5. doi: 10.1111/j.1365-3156.2012.02982.x. Epub 2012 Apr 5. PMID 22487689
- [Result] Alvarez-Uria G, Midde M, Pakam R, Kannan S, Bachu L, Naik PK. Factors Associated with Late Presentation of HIV and Estimation of Antiretroviral Treatment Need according to CD4 Lymphocyte Count in a Resource-Limited Setting: Data from an HIV Cohort Study in India. Interdiscip Perspect Infect Dis. 2012;2012:293795. doi: 10.1155/2012/293795. Epub 2012 Apr 24. PMID 22611389
- [Result] Alvarez-Uria G, Midde M, Pakam R, Bachu L, Naik PK. Effect of Formula Feeding and Breastfeeding on Child Growth, Infant Mortality, and HIV Transmission in Children Born to HIV-Infected Pregnant Women Who Received Triple Antiretroviral Therapy in a Resource-Limited Setting: Data from an HIV Cohort Study in India. ISRN Pediatr. 2012;2012:763591. doi: 10.5402/2012/763591. Epub 2012 Jun 3. PMID 22701801
- [Result] Revell AD, Wang D, Wood R, Morrow C, Tempelman H, Hamers RL, Reiss P, van Sighem AI, Nelson M, Montaner JS, Lane HC, Larder BA; RDI Data and Study Group. An update to the HIV-TRePS system: the development and evaluation of new global and local computational models to predict HIV treatment outcomes, with or without a genotype. J Antimicrob Chemother. 2016 Oct;71(10):2928-37. doi: 10.1093/jac/dkw217. Epub 2016 Jun 20. PMID 27330070
- [Result] Alvarez-Uria G, Midde M, Naik PK. Mortality in HIV-infected patients with tuberculosis treated with streptomycin and a two-week intensified regimen: data from an HIV cohort study using inverse probability of treatment weighting. PeerJ. 2016 May 17;4:e2053. doi: 10.7717/peerj.2053. eCollection 2016. PMID 27231666
- [Result] Alvarez-Uria G, Midde M, Pakam R, Yalla PS, Naik PK, Reddy R. Short-Course Induction Treatment with Intrathecal Amphotericin B Lipid Emulsion for HIV Infected Patients with Cryptococcal Meningitis. J Trop Med. 2015;2015:864271. doi: 10.1155/2015/864271. Epub 2015 Sep 10. PMID 26448766
- [Result] Alvarez-Uria G, Pakam R, Midde M, Yalla PS, Naik PK. Adding Streptomycin to an Intensified Regimen for Tuberculous Meningitis Improves Survival in HIV-Infected Patients. Interdiscip Perspect Infect Dis. 2015;2015:535134. doi: 10.1155/2015/535134. Epub 2015 Aug 4. PMID 26347376
- [Result] Alvarez-Uria G, Pakam R, Midde M, Naik PK. Incidence and mortality of tuberculosis before and after initiation of antiretroviral therapy: an HIV cohort study in India. J Int AIDS Soc. 2014 Dec 9;17(1):19251. doi: 10.7448/IAS.17.1.19251. eCollection 2014. PMID 25499123
- [Result] Alvarez-Uria G, Pakam R, Naik PK, Midde M. Induction with lopinavir-based treatment followed by switch to nevirapine-based regimen versus non-nucleoside reverse transcriptase inhibitors-based treatment for first line antiretroviral therapy in HIV infected children three years and older. PLoS One. 2014 Sep 18;9(9):e108063. doi: 10.1371/journal.pone.0108063. eCollection 2014. PMID 25232730
- [Result] Alvarez-Uria G, Midde M, Pakam R, Naik PK. Directly-observed intermittent therapy versus unsupervised daily regimen during the intensive phase of antituberculosis therapy in HIV infected patients. Biomed Res Int. 2014;2014:937817. doi: 10.1155/2014/937817. Epub 2014 Jun 11. PMID 25013814
- [Result] Alvarez-Uria G, Naik PK, Midde M, Pakam R. Mortality and Loss to Follow up Before Initiation of Antiretroviral Therapy Among HIV-Infected Children Eligible for HIV Treatment. Infect Dis Rep. 2014 May 13;6(2):5167. doi: 10.4081/idr.2014.5167. eCollection 2014 May 13. PMID 25002959
- [Result] Alvarez-Uria G. Description of the cascade of care and factors associated with attrition before and after initiating antiretroviral therapy of HIV infected children in a cohort study in India. PeerJ. 2014 Mar 13;2:e304. doi: 10.7717/peerj.304. eCollection 2014. PMID 24688879
- [Result] Alvarez-Uria G, Naik PK, Midde M, Pakam R. Predictors of loss to follow-up after engagement in care of HIV-infected children ineligible for antiretroviral therapy in an HIV cohort study in India. Germs. 2014 Mar 3;4(1):9-15. doi: 10.11599/germs.2014.1049. eCollection 2014 Mar. PMID 24639956
- [Result] Alvarez-Uria G, Pakam R, Midde M, Naik PK. Optimal Duration of Daily Antituberculosis Therapy before Switching to DOTS Intermittent Therapy to Reduce Mortality in HIV Infected Patients: A Duration-Response Analysis Using Restricted Cubic Splines. Int Sch Res Notices. 2014 Dec 15;2014:704980. doi: 10.1155/2014/704980. eCollection 2014. PMID 27433510
- [Result] Alvarez-Uria G, Naik PK, Midde M, Pakam R. Predictors of delayed entry into medical care of children diagnosed with HIV infection: data from an HIV cohort study in India. ScientificWorldJournal. 2013 Nov 14;2013:737620. doi: 10.1155/2013/737620. eCollection 2013. PMID 24348184
- [Result] Alvarez-Uria G, Pakam R, Midde M, Naik PK. Predictors of delayed antiretroviral therapy initiation, mortality, and loss to followup in HIV infected patients eligible for HIV treatment: data from an HIV cohort study in India. Biomed Res Int. 2013;2013:849042. doi: 10.1155/2013/849042. Epub 2013 Oct 29. PMID 24288689
- [Result] Revell AD, Wang D, Wood R, Morrow C, Tempelman H, Hamers R, Alvarez-Uria G, Streinu-Cercel A, Ene L, Wensing A, Reiss P, van Sighem AI, Nelson M, Emery S, Montaner JS, Lane HC, Larder BA; RDI Study Group. An update to the HIV-TRePS system: the development of new computational models that do not require a genotype to predict HIV treatment outcomes. J Antimicrob Chemother. 2014 Apr;69(4):1104-10. doi: 10.1093/jac/dkt447. Epub 2013 Nov 24. PMID 24275116
- [Result] Revell AD, Alvarez-Uria G, Wang D, Pozniak A, Montaner JS, Lane HC, Larder BA. Potential impact of a free online HIV treatment response prediction system for reducing virological failures and drug costs after antiretroviral therapy failure in a resource-limited setting. Biomed Res Int. 2013;2013:579741. doi: 10.1155/2013/579741. Epub 2013 Sep 24. PMID 24175292
- [Result] Alvarez-Uria G, Midde M, Pakam R, Naik PK. Diagnostic and Prognostic Value of Serum Albumin for Tuberculosis in HIV Infected Patients Eligible for Antiretroviral Therapy: Datafrom an HIV Cohort Study in India. Bioimpacts. 2013;3(3):123-8. doi: 10.5681/bi.2013.025. Epub 2013 Sep 1. PMID 24163804
- [Result] Alvarez-Uria G, Midde M, Pakam R, Naik PK. Predictors of attrition in patients ineligible for antiretroviral therapy after being diagnosed with HIV: data from an HIV cohort study in India. Biomed Res Int. 2013;2013:858023. doi: 10.1155/2013/858023. Epub 2013 Aug 29. PMID 24069604
- [Result] Alvarez-Uria G, Naik PK, Pakam R, Midde M. Factors associated with attrition, mortality, and loss to follow up after antiretroviral therapy initiation: data from an HIV cohort study in India. Glob Health Action. 2013 Sep 12;6:21682. doi: 10.3402/gha.v6i0.21682. PMID 24028937
- [Result] Alvarez-Uria G, Midde M, Pakam R, Naik PK. Initial Antituberculous Regimen with Better Drug Penetration into Cerebrospinal Fluid Reduces Mortality in HIV Infected Patients with Tuberculous Meningitis: Data from an HIV Observational Cohort Study. Tuberc Res Treat. 2013;2013:242604. doi: 10.1155/2013/242604. Epub 2013 Aug 20. PMID 23997952
- [Result] Alvarez-Uria G, Pakam R, Midde M, Naik PK. Entry, Retention, and Virological Suppression in an HIV Cohort Study in India: Description of the Cascade of Care and Implications for Reducing HIV-Related Mortality in Low- and Middle-Income Countries. Interdiscip Perspect Infect Dis. 2013;2013:384805. doi: 10.1155/2013/384805. Epub 2013 Jul 10. PMID 23935613
- [Result] Alvarez-Uria G. Factors associated with delayed entry into HIV medical care after HIV diagnosis in a resource-limited setting: Data from a cohort study in India. PeerJ. 2013 Jun 18;1:e90. doi: 10.7717/peerj.90. Print 2013. PMID 23802091
- [Result] Revell AD, Wang D, Wood R, Morrow C, Tempelman H, Hamers RL, Alvarez-Uria G, Streinu-Cercel A, Ene L, Wensing AM, DeWolf F, Nelson M, Montaner JS, Lane HC, Larder BA; RDI study group. Computational models can predict response to HIV therapy without a genotype and may reduce treatment failure in different resource-limited settings. J Antimicrob Chemother. 2013 Jun;68(6):1406-14. doi: 10.1093/jac/dkt041. Epub 2013 Mar 13. PMID 23485767
- [Result] Alvarez-Uria G, Naik PK, Pakam R, Bachu L, Midde M. Natural History and Factors Associated with Early and Delayed Mortality in HIV-Infected Patients Treated of Tuberculosis under Directly Observed Treatment Short-Course Strategy: A Prospective Cohort Study in India. Interdiscip Perspect Infect Dis. 2012;2012:502012. doi: 10.1155/2012/502012. Epub 2012 Dec 18. PMID 23316226
- [Result] Alvarez-Uria G, Azcona JM, Midde M, Naik PK, Reddy S, Reddy R. Rapid Diagnosis of Pulmonary and Extrapulmonary Tuberculosis in HIV-Infected Patients. Comparison of LED Fluorescent Microscopy and the GeneXpert MTB/RIF Assay in a District Hospital in India. Tuberc Res Treat. 2012;2012:932862. doi: 10.1155/2012/932862. Epub 2012 Aug 26. PMID 22966426
- [Result] Alvarez-Uria G, Midde M, Naik PK. Socio-demographic Risk Factors Associated with HIV Infection In Patients Seeking Medical Advice in a Rural Hospital of India. J Public Health Res. 2012 Feb 14;1(1):79-82. doi: 10.4081/jphr.2012.e14. eCollection 2012 Feb 17. PMID 25170450
- [Result] Alvarez-Uria G, Naik PK, Midde M, Kannan S, Reddy R. False negative HIV antibody test in HIV infected children who receive early antiretroviral treatment in a resource-limited setting. Infect Dis Rep. 2012 Jan 4;4(1):e6. doi: 10.4081/idr.2012.e6. eCollection 2012 Jan 2. PMID 24470936
- [Result] Alvarez-Uria G, Reddy R, Reddy S, Naik PK, Midde M. Evaluation of a Low-Cost Strategy for Enumerating CD4 Lymphocyte Absolute Count and Percentage Using the FACSCalibur Flow Cytometer in HIV-Infected Patients from a Resource-Limited Setting. ISRN AIDS. 2012 Oct 23;2012:494698. doi: 10.5402/2012/494698. eCollection 2012. PMID 24052877
- [Result] Alvarez-Uria G, Midde M, Naik PK. Trends and risk factors for HIV infection among young pregnant women in rural India. Int J Infect Dis. 2012 Feb;16(2):e121-3. doi: 10.1016/j.ijid.2011.10.003. Epub 2011 Dec 5. PMID 22153000